CLINICAL TRIAL: NCT04421612
Title: COVID-19 - No Health Without Mental Health
Acronym: Co-COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 126376
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2020-08

CONDITIONS: Covid19; Anxiety
MeSH Terms: conditions — COVID-19; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Group one recieve a new module every three days. Group two recive a new module every 5 days.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive (Experimental): This group recieve access to a new module every 3rd day.
  Interventions: Behavioral: Co-mestring (co-coping)
- Ordinary (Experimental): This group recieve access to a new module every 5th day.
  Interventions: Behavioral: Co-mestring (co-coping)

INTERVENTIONS:
Behavioral: Co-mestring (co-coping) — 8 modules with the aim to reduce stress, increase coping of social isolation and coping with the consequences of reduced positive experiences

SUMMARY:
The Corona pandemic is affecting the whole world and since March 12.th 2020 there has been strict qurantene and social isolation interventions in Norway. The aim of this intervention is to reduce the negative and fatal effects of the pandemic. The pandemic and the restrictions that follows it is assumed to affect the mental health of the general population. In this research project we want to examine the use and the effects of a digital self-guided psychological intervention with the aim to increase coping and to reduce psychological problems during and after the pandemic. The participants will be randomized to either an intensive group (new module every 3rd day) or to an ordinary group (new module every 5th day).

DETAILED DESCRIPTION:
The intervention was developed in a crossdiciplinary and cross-sectorial team within the framework of the research project INTROMAT, an ICT Lighthouse research project funded by the Norwegian Research Council. The content of the digital covid-19 intervention was based on four previously developed digital interventions, all based on systematic user-involvement and user-testing, from our group. The person-based approach inspired the development of the intervention. Based on the research literature and experience from our existing digital interventions we started the development with establishing guiding principles. The intervention consists of 8 modules.

ELIGIBILITY:
Inclusion Criteria:

* read and write norwegian
* above 18 years
* Mild and moderate stress

Exclusion Criteria:

* current treatment for mental health disorders
* history or present severe mental health disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
The Patient Health Questionnaire | 6 months
  measures depression severity with nine items scored 0 ("not at all") to 3 ("nearly every day"), corresponding to the criteria for major depression in the DSM-5. The sum of the scores for the nine items ranges from 0 to 27
The Generalized Anxiety Disorder Scale | 6 months
  measures anxiety severity with seven items scored 0 ("not at all") to 3 ("nearly every day"). The total score ranges from 0 to 21

SECONDARY OUTCOMES:
Positive and negative affect | 6 months
  In the instructions to the PANAS scales in the current study, participants were asked, ''To what extent do you generally feel this way, that is, how do you feel on average?'' Each PANAS scale comprises 10 specific mood-related adjectives, rated on a 5-point scale from not at all to very much
Perceived Stress Scale | 6 months
  Widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives.
Client Satisfaction Scale | 6 months
  structured survey used to assess level of satisfaction with care. Items are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction) with different descriptors for each response point. Total scores range from 8 to 32, with higher scores indicating greater satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided
There is a plan to share anonymous interaction-data. Health data are undecided